CLINICAL TRIAL: NCT04762017
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of OCS-05 in Patients With Acute Optic Neuritis
Brief Title: OCS-05 in Patients With Optic Neuritis
Acronym: ACUITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oculis (Industry)
Collaborators: Neurotrials (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OCS-05_P2_01; 2020-003147-29 (EudraCT Number)
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Optic Neuritis
Keywords: Acute Optic Neuritis (AON); Optic Neuritis
MeSH Terms: conditions — Optic Neuritis | interventions — Adrenal Cortex Hormones; Organization and Administration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCS-05 +SoC (corticosteroid IV) (Experimental): Once daily IV infusions of OCS-05 + SoC (corticosteroid) (n=18) for 5 consecutive days
  Interventions: Drug: OCS-05 +SoC (corticosteroid) IV administration
- Placebo +SoC (corticosteroid IV) (Placebo Comparator): Once daily IV infusions of Placebo + SoC (corticosteroid) (n=18) for 5 consecutive days
  Interventions: Other: Placebo + SoC (corticosteroid) IV administration

INTERVENTIONS:
Drug: OCS-05 +SoC (corticosteroid) IV administration — OCS-05 + SoC (corticosteroid) IV administration for 5 consecutive days
  Arms: OCS-05 +SoC (corticosteroid IV)
Other: Placebo + SoC (corticosteroid) IV administration — Placebo + SoC (corticosteroid) IV administration for 5 consecutive days
  Arms: Placebo +SoC (corticosteroid IV)

SUMMARY:
To evaluate the safety and tolerability of OCS-05 compared to placebo in patients with optic neuritis receiving the standard of care

DETAILED DESCRIPTION:
ACUITY is a phase 2, multicentric, two-arm, randomized, double-blind, placebo-controlled study to evaluate the safety and tolerability of OCS-05 compared to placebo in patients with acute optic neuritis (AON) receiving the standard of care. Patients received OCS-05 2mg/kg/day, 3mg/kg/day or placebo for five days in addition corticosteroid standard of care (SoC).

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosed with a unilateral optic neuritis
* Onset of visual loss symptoms in the last 12 days before randomization

Main Exclusion Criteria:

* Optic neuropathy of non-demyelinating origin
* Known Neuromyelitis optica with autoantibodies against aquaporin-4 (AQP4-Abs)
* Patients with widespread and symmetric white matter alterations in the screening MRI suggestive of other demyelinating disorders (e.g. metabolic disorders, mitochondrial disorders)
* Active, chronic disease (or stable but treated with immune therapy) of the immune system other than Multiple Sclerosis (MS) or Myelin Oligodendrocyte Glycoprotein Antibody associated Disorder (MOGAD)(e.g. Sjögren's disease, systemic lupus erythematosus) or with a known immunodeficiency syndrome (AIDS, hereditary immune deficiency, drug induced immune deficiency)
* An alternative cause of visual loss (e.g. compressive or infiltrative lesion of the optic nerve, infections, genetic forms of visual loss.
* Diagnosed with macular edema, severe myopia (>6 δ) or other disease of the retina at inclusion
* Known diabetic retinopathy
* Known glaucoma
* Female patients of child-bearing potential who are unwilling to use an effective contraception while enrolled on study and for the duration of the study.
* Male patients not willing to use contraception (abstinence, condom etc..) while enrolled in the study and receiving the experimental drug, and for at least 2 days after the last experimental drug administration.
* Breastfeeding or pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with shift from normal (baseline) to abnormal in ECG parameters. | From Day 1 (V3-t1 after investigational drug administration) to Day 15 (V4)
  To determine the shift from normal to abnormal ECG parameters.

SECONDARY OUTCOMES:
Describe the Ganglion Cell and Inner Plexiform Layer (GCIPL) thickness, absolute and relative change from baseline (of the affected eye) to each time point (t5, M1, M3, M6) | Up to 6 months
  To determine the change in retinal layers thickness from baseline in the affected eye
Describe the Retinal Nerve Fiber Layer (RNFL) thickness, absolute and relative change from baseline (of the affected eye) to each time point (t5, M1, M3, M6). | Up to 6 months
  To determine the change in retinal layers thickness from baseline in the affected eye.
To describe the visual function on the 2.5% ETDRS Low Contrast Letter Acuity (LCVA) chart change from baseline (of the affected eye) to each time point (D15, M1, M3, M6) | Up to 6 months
  To determine change in clinical vision parameters in the affected eye as compared to baseline.
To describe the visual function on the 2.5% ETDRS High Contrast Letter Acuity (HCVA) chart change from baseline (of the affected eye) to each time point (D15, M1, M3, M6) | Up to 6 months
  Change in clinical vision parameters in the affected eye as compared to baseline
To describe the visual function on the Humphrey visual fields evaluations change from baseline (of the affected eye) to each time point (M1, M3, M6) | Up to 6 months
  Change in clinical vision parameters in the affected eye as compared to baseline
To summarize the Visual Evoked Potential latency and amplitude and the change from baseline of the affected eye to each time point (M3 and M6) by treatment group and OCS-05 pooled group | Up to 6 months
  Change in electrophysiological parameters in the affected eye as compared to baseline
To summarize the EDSS (Expanded Disability Status Scale) scores and the change from baseline to each time point (M1, M3 and M6) by treatment group and OCS-05 pooled group | Up to 6 months
  Change in neurological parameters in the affected eye as compared to baseline
To describe the rate of treatment switch at 6 months for subjects receiving Disease Modifying Therapy (DMT) for multiple sclerosis | 6 months
  Change in rate of treatment switch for subjects receiving Disease Modifying Therapy (DMT) for multiple sclerosis
To summarize the incidence of safety parameters including clinically notable laboratory abnormalities | Up to 6 months
  Change in safety laboratory parameters as compared to baseline
To describe the Cmax of OCS-05 for patients having the full PK scheme and for patients having the single PK point at 1.5h post infusion on Day 1 | Day 1
  Characterize the PK profile of OCS-05 3mg/kg
To describe the Tmax of OCS-05 for patients having the full PK scheme and for patients having the single PK point at 1.5h post infusion on Day 1 | Day 1
  Characterize the PK profile of OCS-05 3mg/kg
To describe the AUC0-t of OCS-05 for patients having the full PK scheme and for patients having the single PK point at 1.5h post infusion on Day 1 | Day 1
  Characterize the PK profile of OCS-05 3mg/kg

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Klier, MD, MPH, Study Director — Oculis
Locations (4):
- France (4):
  - Hospices Civils de Lyon, Lyon
  - CHU - Nice, Nice
  - CIC Neurosciences - La Pitié Salpêtrière, Paris
  - Foundation Rothschild, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villoslada P, Masso M, Paris S, Hutchings S, Koch A. A Phase 1 randomized study on the safety and pharmacokinetics of OCS-05, a neuroprotective disease modifying treatment for Acute Optic Neuritis and Multiple Sclerosis. Sci Rep. 2023 Mar 29;13(1):5099. doi: 10.1038/s41598-023-32278-0. PMID 36991169